CLINICAL TRIAL: NCT05594992
Title: An Extension Study of JR-141 to Evaluate the Long-term Safety and Efficacy in Mucopolysaccharidosis Type II (Hunter Syndrome) Subjects
Brief Title: An Extension Study of JR-141 to Evaluate the Long-term Safety and Efficacy in MPS II (Hunter Syndrome) Subjects
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JR-141-GS32
Record Dates: First submitted 2022-10-06; First posted 2022-10-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Mucopolysaccharidosis II
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JR-141 2.0 mg/kg/week (Experimental)
  Interventions: Drug: JR-141

INTERVENTIONS:
Drug: JR-141 — IV infusion, 2.0 mg/kg/week

SUMMARY:
An extension of Global Phase III open-label, multicenter designed to evaluate the Long-term safety and efficacy of study drug for the treatment of the MPS II.

ELIGIBILITY:
Inclusion Criteria:

1. A subject who participated in the Parent Study (JR-141-GS31) and completed the assessments at Week 105 in Cohort A or Week 53 in Cohort B before being administered the study medication of that respective visit, and in the opinion of the principal investigator there are no safety concerns.
2. A subject from whom an IRB or IEC-approved written informed consent can be obtained, which is voluntarily signed. If the subject is aged under 18 years (aged under 16 years in the UK) at the time of enrollment or willingness to participate in the study cannot be confirmed due to MPS II-related intellectual disability, the subject's legally acceptable representative (e.g., his parents or guardians) may sign the ICF on behalf of the subject. Written informed assent should be obtained from the subject, wherever possible.
3. Female subject of child bearing potential or male subject whose female partner is of child-bearing potential, i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile, agrees to use a medically accepted, highly effective method of contraception from the time of signing the ICF. The method of contraception must be used during the study until 90 days for male subjects, and 30 days for female subjects after the final study drug administration.

Exclusion Criteria:

1. A subject who changed treatment from JR-141 to idursulfase during the treatment period in the Parent Study (JR-141-GS31).
2. A subject who is unable to comply with the protocol (e.g., is unable to return for safety evaluations or is otherwise unlikely to complete the study) as determined by the principal investigator or sub-investigator.
3. [Only in France] Persons deprived of their liberty by a judicial or administrative decision, according to article L. 1121-6 of the Public Health Code (Code de la santé publique, CSP) adults who are the subject of a measure of legal protection or unable to express their consent according to article L. 1121-8 of the CSP.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in heparan sulfate concentrations in cerebrospinal fluid from each subject's first administration of JR-141 throughout the Parent Study (JR-141-GS31) or this study to each time point | [A-1, A-2, A-3: Week 157, 209, 261] [A-4: Week 131, 183, 235, 287]
  Assessment will be mandatory for the first two years after starting JR-141 administration through the parent study or the extension study.
Change in neurocognitive testing, calculated by the BSID-III or KABC-II, from each subject's first administration of JR-141 throughout the Parent Study (JR-141-GS31) or this study | [A-1: Week 157, 209, 261] [A-2: Week 131, 157, 183, 209, 261] [A-3: Week 131, 157, 209, 261 ] [A-4: Week 131, 157, 183, 235, 287]
Change in neurocognitive testing, calculated by the VABS-II from each subject's first administration of JR-141 throughout the Parent Study (JR-141-GS31) or this study | [A-1: Week 157, 209, 261] [A-2: Week 131, 157, 183, 209, 261] [A-3: Week 131, 157, 209, 261 ] [A-4: Week 131, 157, 183, 235, 287][B-1: Week 78, 105, 157, 209, 261] [B-2: Week 78, 105, 131, 157, 209, 261]
Change in neurocognitive testing, calculated by the Wechsler, from each subject's first administration of JR-141 throughout the Parent Study (JR-141-GS31) or this study | [B-1: Week 78, 105, 157, 209, 261] [B-2: Week 78, 105, 131, 157, 209, 261]

SECONDARY OUTCOMES:
Change in liver and spleen volume from each subject's first administration of JR-141 throughout the Parent Study (JR-141-GS31) or this study | [A-1, A-3: Week 157, 209, 261] [A-2: Week 131, 157, 209, 261] [A-4: Week 131, 183, 235, 287] [B-1: Week 105, 157, 209, 261] [B-2: Week 78, 105, 157, 209, 261]
Change in 6-minute walk distance from each subject's first administration of JR-141 throughout the Parent Study (JR-141-GS31) or this study | [B-1: Week 105, 157, 209, 261] [B-2: Week 78, 105, 157, 209, 261]

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hospital Universitario Austral, Buenos Aires, Argentina
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Instituto de Genética e Erros Inatos do Metabolismo, São Paulo
- Hôpital Femme Mère Enfant, Bron, France
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Osp. Pediatrico Bambino Gesù, IRCCS, Rome, Italy
- Uniwersytecki Szpital Dziecięcy, Krakow, Poland
- Hospital Sant Joan de Déu, Barcelona, Spain